CLINICAL TRIAL: NCT06490549
Title: An Epidemiological Study to Investigate the Characteristics of RSV Infection in Adult Hematopoietic Cell Transplant Recipients or Hematological Malignancies Patients in Tianjin HI (Hematology Institute)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Other Study IDs: IIT2023069
Record Dates: First submitted 2023-12-06; First posted 2024-07-08 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2023-12

CONDITIONS: RSV Infection
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: RSV infection observation cohort — No intervention; Epidemiological Study. Participants will receive standard care based on local clinical practice

SUMMARY:
This primary objective of this study is to describe the incidence of RSV infection in adult hematopoietic cell transplant recipients OR hematological malignancies patients in Tianjin HI.

ELIGIBILITY:
Inclusion Criteria:

* 1) Aged ≥ 18 years old. 2) Receiving hematopoietic stem cell transplantation; OR being diagnosed with hematological malignancies (including but not limited to leukemia, lymphoma, and multiple myeloma) and receiving chemotherapy.

  3) New onset of respiratory symptoms; OR exacerbation of existing chronic respiratory symptoms (such as previously diagnosed chronic runny nose, seasonal allergies, chronic lung disease, etc.).

  4) Willing to sign an informed consent form, able to understand and willing to follow the study protocol.

Exclusion Criteria:

* Unwillingness to sign an informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult hematopoietic stem cell transplantation (HCT) recipients OR hematological malignancies (HM) patients have new onset or worsen of respiratory signs/syndromes and presented the study site.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-11-30 (Actual); Primary Completion 2025-06-20 (Estimated); Study Completion 2025-06-20 (Estimated)

PRIMARY OUTCOMES:
the incidence of RSV infection in adult hematopoietic stem cell transplantation (HCT) recipients OR hematological malignancies (HM) patients presenting the study site | 1 year
  infection incidence
the Incidence of RSV infection in adult hematopoietic stem cell transplantation (HCT) recipients OR hematological malignancies (HM) patients presenting the hospital | 1 year
  infection incidence

SECONDARY OUTCOMES:
the clinical characteristics of RSV infection | 1 year
  symptoms description and scoring of RSV infection
Clinical outcome and relevant risk factor of RSV infection | 1 year
  Clinical outcome and relevant risk factor of RSV infection
Virological characteristics of RSV infection from D1 through D28, D42 or even longer | 1 year
  Clinical outcome and relevant risk factor of RSV infection

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Chinese Academy of Medical Sciences, Tianjin, China

IPD SHARING:
Plan to Share IPD: No